CLINICAL TRIAL: NCT05502510
Title: Assessing the Effectiveness and Efficacy of the MyHealthyPregnancy Application
Status: Completed | Type: Observational
Sponsor: Naima Health LLC (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Sponsor
Other Study IDs: 1684
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy Related; Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MyHealthyPregnancy (MHP): Use of the MyHealthyPregnancy application in conjunction with usual care.
  Interventions: Behavioral: MyHealthyPregnancy
- Usual Prenatal Care (usual care): Usual prenatal care consisting of biweekly visits with the patient care team.

INTERVENTIONS:
Behavioral: MyHealthyPregnancy — MyHealthyPregnancy is a mobile application prescribed to expectant mothers in conjunction with normal prenatal care. The application uses behavioral decision science principles to identify risks of preterm birth and alert the mother and care team of these risks.
  Groups: MyHealthyPregnancy (MHP)

SUMMARY:
One in ten births will occur prior to 37 weeks of gestation leading to serious complications such as problems with lung, heart and brain function and an increased risk of infant mortality. Solutions exist to treat risk factors related to preterm birth but these solutions require timely identification of the risks which is often not possible within regular prenatal care. This study will evaluate MyHealthyPregnancy, an application that monitors for common risks associated with preterm birth and recommends solutions to the expectant mother and care team.

DETAILED DESCRIPTION:
MyHealthyPregnancy (MHP) is an application that was developed using behavioral decision science principles. This study seeks to evaluate the effectiveness and efficacy of the application. MyHealthyPregnancy was offered to expectant mothers at the University of Pittsburgh Medical Center in conjunction with usual prenatal care. The primary objective is to compare the reduction in gestational age at birth between MHP and usual care cohorts. Secondary objectives include comparing births occurring prior to 37 weeks of gestation, depression rates, anxiety rates, referrals to behavioral health, referrals to social workers, preeclampsia rates, gestational weight gain, number of prenatal appointments attended, and percent of required prenatal appointments attended between the MHP and usual care cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Offered a prescription for MyHealthyPregnancy
* 18+ years of age
* Pregnant
* Seeking care at a UPMC hospital
* Delivered at a UPMC hospital

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant people offered a prescription for MyHealthyPregnancy who were at least 18 years of age, pregnant, received care at UPMC, and delivered at a UPMC hospital
Sampling Method: Non-Probability Sample
Enrollment: 12344 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Gestational Age at Birth | Baseline to 40 Weeks
  Gestational age at birth will be measured using each patients electronic health record. The average treatment effect will be calculated using linear regression comparing MHP and usual care cohorts.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects gestational age at birth.

SECONDARY OUTCOMES:
Prenatal Births | Baseline to 37 Weeks
  Occurrence of preterm birth will be measured using each patient's electronic health record. The likelihood of preterm birth between the MHP and usual care cohorts will be compared using logistic regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects preterm birth.
Depression Rates | Baseline to 40 Weeks
  Depression rates will be measured using diagnoses of depression in each patient's electronic health record. Depression rates between the MHP and usual care cohorts will be compared using linear regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects depression rates.
Anxiety Rates | Baseline to 40 Weeks
  Anxiety rates will be measured using diagnoses of anxiety in each patient's electronic health record. Anxiety rates between the MHP and usual care cohorts will be compared using linear regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects anxiety rates.
Referrals to Behavioral Health Specialists | Baseline to 40 Weeks
  Rates of referrals to behavioral health specialists will be measured using each patient's electronic health record. Rates in referrals between the MHP and usual care cohorts will be compared using linear regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects rates of referrals.
Referrals to Social Workers | Baseline to 40 Weeks
  Rates of referrals to social workers will be measured using each patient's electronic health record. Rates in referrals between the MHP and usual care cohorts will be compared using linear regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects rates of referrals.
Preeclampsia | Baseline to 40 Weeks
  Preeclampsia will be measured using each patient's electronic health record. Rates of preeclampsia between the MHP and usual care cohorts will be compared using linear regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects preeclampsia.
Gestational Weight Gain | Baseline to 40 Weeks
  Gestational weight gain will be measured by calculating the difference between each patient's initial weight and delivery weight recorded in their electronic health record. Gestational weight gain will be categorized as sufficient or insufficient according to 2009 Institute of Medicine guidelines. The likelihood of achieving sufficient gestational weight gain between the MHP and usual care cohorts will be compared using ordinal regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects the likelihood of achieving sufficient gestational weight gain.
Attendance at Prenatal Appointments | Baseline to 40 Weeks
  Number of prenatal visits attended will be measured using each patient's electronic health record. The number of visits attended between the MHP and usual care cohorts will be compared using linear regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects attendance at prenatal visits.
Attendance at Required Prenatal Appointments | Baseline to 40 Weeks
  The percent of required prenatal appointments attended will be measured using each patient's electronic health record. The percent of visits attended between the MHP and usual care cohorts will be compared using linear regression.
  Efficacy of the application will be assessed using a dose-response model to evaluate how use of the application affects attendance at prenatal visits.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Analytic Code — https://osf.io/bty8n/?view_only=f8bb6e5a7698443494d4c3788a45cc0f — The analytic code will be uploaded to OSF upon publishing the manuscript.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT05502510/SAP_000.pdf